CLINICAL TRIAL: NCT05160597
Title: Evaluation of 68Ga-PSMA-11 PET Guided Prostate Biopsy in Men With Suspicion of Clinically Significant Prostate Cancer and Prior Negative/Inconclusive Biopsy: A Prospective Exploratory Study
Brief Title: Image-Guided (68Ga-PSMA-11 PET/CT) Prostate Biopsy for the Diagnosis of Prostate Cancer in Men With Prior Negative/Inconclusive Biopsy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-001122; NCI-2021-12975 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-15; First posted 2021-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (68Ga-PSMA-11, image-guided prostate biopsy) (Experimental): SCREENING PROCEDURE: Patients receive 68Ga-PSMA-11 IV and 50-100 minutes later, undergo a PET/CT scan. Only patients with 68Ga-PSMA-11 uptake within the prostate proceed to image-guided biopsy.
  IMAGE-GUIDED BIOPSY: Patients undergo experimental image-guided prostate biopsy using PET/CT images obtained during screening procedure during a standard of care TRUS.
  Interventions: Procedure: Biopsy of Prostate; Other: Gallium Ga 68 Gozetotide; Procedure: Transrectal Ultrasonography Guided Biopsy

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo image-guided prostate biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Transrectal Ultrasonography Guided Biopsy — Undergo standard of care TRUS
  Other Names: TRUS Biopsy; TRUS-Guided Biopsy

SUMMARY:
This early phase I trial studies how well an image-guided prostate biopsy using the imaging agent 68Ga-prostate-specific membrane antigen (PSMA)-11 with a positron emission tomography/computed tomography (PET/CT) scan works in diagnosing prostate cancer in men with a prior negative or inconclusive prostate biopsy. PSMA is a protein that is found on the surface of prostate cancer cells. 68Ga-PSMA-11 is made up of a substance that binds to PSMA on tumor cells, linked with a radioactive substance that can then be seen on imaging scans such as PET/CT. 68Ga-PSMA-11 PET/CT-guided biopsy may help improve the detection rate of prostate cancer. This may help reduce over-diagnosis and over-treatment in men with low-risk prostate cancer and under-treatment in men with high-risk prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the detection rate of clinically significant prostate cancer (Gleason score 7 or more) in patients with focal gallium Ga 68 gozetotide (68Ga-PSMA-11) uptake within the prostate.

OUTLINE:

SCREENING PROCEDURE: Patients receive 68Ga-PSMA-11 intravenously (IV) and 50-100 minutes later, undergo a PET/CT scan. Only patients with 68Ga-PSMA-11 uptake within the prostate proceed to image-guided biopsy.

IMAGE-GUIDED BIOPSY: Patients undergo experimental image-guided prostate biopsy using PET/CT images obtained during screening procedure during a standard of care transrectal ultrasonography guided biopsy (TRUS).

ELIGIBILITY:
Inclusion Criteria:

* Men with suspicion of clinically significant prostate cancer with prior inconclusive, discordant or negative magnetic resonance imaging/ultrasound (MRI/US) fusion prostate biopsy
* Scheduled for a repeat transrectal ultrasound (TRUS) prostate biopsy by standard of care
* Focal 68Ga-PSMA-11 uptake within the prostate

Exclusion Criteria:

* Negative 68Ga-PSMA-11 uptake within the prostate (screening failure)
* Age < 18 and > 90 years
* Recurrent prostate cancer
* Inability to provide written informed consent
* Known inability to remain still and lie flat for the duration of the PET/CT (about 30 minutes)

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Detection rate of clinically significant prostate cancer | Up to 3 years
  Defined as the percentage of clinically significant prostate cancer (Gleason score 7 or more) in patients with focal 68Ga-PSMA-11 uptake within the prostate

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States